CLINICAL TRIAL: NCT00066807
Title: A Phase III Trial Evaluating the Role of Chemotherapy as Adjuvant Therapy for Premenopausal Women With Endocrine Responsive Breast Cancer Who Receive Endocrine Therapy
Brief Title: Premenopausal Endocrine Responsive Chemotherapy Trial
Acronym: PERCHE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual, patients were followed until completion of 5 yrs treatment
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 26-02 / BIG 4-02; NABCI-IBCSG-26-02 (International Breast Cancer Study Group); EU-20401 (Breast International Group); 2005-002626-59 (EudraCT Number); CDR0000318832 (Registry Identifier: CT.gov)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Epirubicin; exemestane; Tamoxifen; Triptorelin Pamoate; Gonadotropin-Releasing Hormone; Ovariectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFS plus T or E (Experimental): Ovarian function suppression (OFS) by triptorelin for 5 years or surgical oophorectomy or ovarian irradiation PLUS tamoxifen (T) or exemestane (E) for 5 years.
  Interventions: Drug: exemestane; Drug: tamoxifen; Drug: triptorelin; Procedure: oophorectomy; Procedure: ovarian irradiation
- Chemotherapy plus OFS plus T or E (Experimental): Chemotherapy plus ovarian function suppression (OFS) by triptorelin for 5 years or surgical oophorectomy or ovarian irradiation PLUS tamoxifen (T) or exemestane (E) for 5 years.
  Interventions: Drug: chemotherapy; Drug: exemestane; Drug: tamoxifen; Drug: triptorelin; Procedure: oophorectomy; Procedure: ovarian irradiation

INTERVENTIONS:
Drug: chemotherapy — Planned duration of chemotherapy: 2 months if an anthracycline is included (e.g., 4 cycles of EC or AC) or 4 months if no anthracycline is given (e.g., 6 cycles of CMF) is recommended. Unless medically contraindicated, an anthracycline-containing regimen using epirubicin should be given.
  Other Names: Ellence; Epirubicin Ebewe
  Arms: Chemotherapy plus OFS plus T or E
Drug: exemestane — Exemestane 25 mg orally daily for until 5 years from date of randomization, unless relapse or intolerance should occur earlier.
  Other Names: Aromasin
Drug: tamoxifen — Tamoxifen 20 mg orally daily until 5 years from date of randomization, unless relapse or intolerance should occur earlier.
  Other Names: Nolvadex
Drug: triptorelin — Triptorelin (GnRH analogue) 3.75 mg by intramuscular injection every 28 days for 5 years from randomization, unless relapse or intolerance should occur earlier or surgical oophorectomy or ovarian irradiation is subsequently performed.
  Other Names: GnRH analog; Trelstar Depot
Procedure: oophorectomy — Bilateral surgical oophorectomy via laparotomy or laparoscopy.
Procedure: ovarian irradiation — Bilateral ovarian irradiation.

SUMMARY:
The PERCHE trial evaluated the worth of adding adjuvant chemotherapy for premenopausal women with steroid hormone receptor positive early invasive breast cancer who receive ovarian function suppression plus either tamoxifen or exemestane for five years. The use of chemotherapy was determined by randomization. The method of ovarian function suppression (GnRH analogue for five years, surgical oophorectomy or ovarian irradiation) and the choice of tamoxifen or exemestane were determined by the investigator or by randomization in the IBCSG 25-02 TEXT trial [recommended option]. The trial was terminated early due to poor accrual.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare ovarian function suppression and tamoxifen or exemestane with vs without adjuvant chemotherapy in premenopausal women with endocrine-responsive resected breast cancer.
* Compare the disease-free and overall survival of patients treated with these regimens.
* Compare sites of first treatment failure in patients treated with these regimens.
* Compare the incidence of second nonbreast malignancies in patients treated with these regimens.
* Compare the quality of life, including late side effects of early menopause, of patients treated with these regimens.

PLANNED OUTLINE:

This is a randomized, multicenter study. Patients are stratified according to participating center, number of positive axillary and/or internal mammary lymph nodes (0 vs 1 or more), method of ovarian function suppression (triptorelin vs oophorectomy vs ovarian irradiation), chemotherapy if randomized to arm II (not containing vs containing an anthracycline or taxane), and endocrine agent (tamoxifen vs exemestane vs selected by subsequent randomization in the TEXT trial). Treatment duration is five years.

Quality of life is assessed at baseline, every 6 months for 2 years, and then annually for 4 years. Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter.

NOTE: Trial was terminated early due to poor accrual.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer confined to the breast and axillary nodes

  * No distant metastatic disease
  * Tumor detected in the internal mammary chain by sentinel node procedure allowed
* Must have undergone 1 of the following procedures for primary breast cancer within the past 12 weeks and have no known clinical residual locoregional disease:

  * Total mastectomy with or without adjuvant radiotherapy
  * Breast-conserving surgery (e.g., lumpectomy, quadrantectomy, or partial mastectomy with margins clear* of invasive cancer and ductal carcinoma in situ) followed by radiotherapy NOTE: *If all other margins are clear, a positive posterior (deep) margin is permitted, provided the excision was performed down to the pectoral fascia and all tumor has been removed OR a positive anterior (superficial; abutting skin) margin is allowed provided all tumor was removed
* Prior axillary lymph node dissection or negative axillary sentinel node biopsy required

  * Patients with microscopically positive axillary sentinel nodes allowed provided they were evaluated on a clinical trial evaluating microscopically positive lymph nodes
* No locally advanced, inoperable breast cancer, including any of the following characteristics:

  * Inflammatory breast cancer
  * Supraclavicular node involvement
  * Enlarged internal mammary nodes (unless pathologically negative)
* No prior ipsilateral or contralateral invasive breast cancer

  * Histologically diagnosed synchronous bilateral invasive breast cancer within the past 2 months allowed if the bilateral disease meets all other eligibility criteria
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor positive in each tumor

    * At least 10% of tumor cells positive by immunohistochemistry

PATIENT CHARACTERISTICS:

Age

* Premenopausal

Sex

* Female

Menopausal status

* Premenopausal

  * Estradiol in the premenopausal range after surgery

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No systemic hepatic disease that would preclude prolonged follow-up

Renal

* No systemic renal disease that would preclude prolonged follow-up

Cardiovascular

* No prior deep venous thrombosis and/or embolism unless patient is medically suitable
* No systemic cardiovascular disease that would preclude prolonged follow-up

Pulmonary

* No systemic pulmonary disease that would preclude prolonged follow-up

Other

* Not pregnant or nursing
* Fertile patients must use effective nonhormonal contraception
* No other prior or concurrent invasive malignancy except adequately treated basal cell or squamous cell skin cancer, nonbreast carcinoma in situ without invasion, contralateral or ipsilateral carcinoma in situ of the breast
* No prior or concurrent nonbreast invasive malignancy within the past 5 years that is nonrecurrent including any of the following:

  * Stage I papillary thyroid cancer
  * Stage Ia carcinoma of the cervix
  * Stage Ia or b endometrioid endometrial cancer
  * Borderline or stage I ovarian cancer
* No other nonmalignant systemic disease that would preclude prolonged follow-up
* No history of noncompliance with medical regimens
* No psychiatric, addictive, or other disorder that would preclude study compliance or giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior neoadjuvant or adjuvant chemotherapy

  * Neoadjuvant or adjuvant trastuzumab (Herceptin®) allowed

Endocrine therapy

* No prior neoadjuvant or adjuvant endocrine therapy after breast cancer diagnosis
* No prior tamoxifen or other selective estrogen-receptor modulator (e.g., raloxifene) within 1 year before the breast cancer diagnosis
* No other concurrent oral or transdermal hormonal therapy, including any of the following:

  * Estrogen
  * Progesterone
  * Androgens
  * Aromatase inhibitors
  * Hormone replacement therapy
  * Oral or other hormonal contraceptives, including implant and depot injections
  * Raloxifene or other selective estrogen-receptor modulators

Radiotherapy

* See Disease Characteristics
* No prior ovarian irradiation

Surgery

* See Disease Characteristics
* No prior bilateral oophorectomy

Other

* No other prior neoadjuvant therapy
* No other concurrent investigational agents
* No concurrent bisphosphonates unless bone density has been documented at least 1.5 standard deviations below the young adult normal mean or the patient is participating in a randomized clinical trial setting testing bisphosphonates in the adjuvant breast cancer setting

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Torrisi, MD, Study Chair — Breast International Group, European Institute of Oncology, Milano, Italy; Edith A. Perez, MD, Study Chair — North American Intergroup, Mayo Clinic Jacksonville, Jacksonville, USA
Locations (6):
- National Institute of Oncology, Budapest, Hungary
- Italy (2):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - European Institute of Oncology, Milan
- Switzerland (3):
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen

REFERENCES:
- [Background] Francis P, Fleming G, Nasi ML, et al.: Tailored treatment investigations for premenopausal women with endocrine responsive (ER+ and/or PGR+) breast cancer: the SOFT, TEXT, and PERCHE trials. [Abstract] The Breast 12 (Suppl 1): A-P104, S44, 2003.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened 4Aug03; the first patient was randomized on 1Jun04. The accrual goal for the study was 1750 patients. A total of 29 patients were randomized as of 31Dec06 when the trial was terminated. 25 of these 29 patients were also enrolled in the TEXT trial (IBCSG 25-02).
Groups:
- OFS Plus T or E for 5 Years: Ovarian function suppression (OFS) by triptorelin for 5 years or surgical oophorectomy or ovarian irradiation PLUS tamoxifen (T) or exemestane (E) for 5 years.
- Chemotherapy Plus OFS Plus T or E for 5 Years: Chemotherapy plus ovarian function suppression (OFS) by triptorelin for 5 years or surgical oophorectomy or ovarian irradiation PLUS tamoxifen (T) or exemestane (E) for 5 years.
Period: Overall Study
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years
Started | 14 | 15
Completed | 0 | 0
Not Completed | 14 | 15
Not completed — Study was terminated early | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 45 [42 to 48] | 45 [42 to 48] | 45 [42 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Time Frame: For first time at a median follow up approximately 5 years
Population: The trial was terminated early due to poor accrual. No outcome measure data is available.
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival
Time Frame: For first time at a median follow up approximately 5 years
Population: The trial was terminated early due to poor accrual. No outcome measure data is available.
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Systemic Disease-free Survival
Time Frame: For first time at a median follow up approximately 5 years
Population: The trial was terminated early due to poor accrual. No outcome measure data is available.
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Sites of First Treatment Failure
Time Frame: For first time at a median follow up approximately 5 years
Population: The trial was terminated early due to poor accrual. No outcome measure data is available.
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5-year protocol treatment period
Description: CAVEAT: Trial was terminated early; data available ONLY for selected Grade 3-5 adverse events for chemotherapy arm. Systematic assessment included form with specific AEs related to chemotherapy. 25 out of 29 patients were co-enrolled in TEXT (IBCSG 25-02) and AEs associated with endocrine therapy are reported as part of that trial.
Arm/Group | OFS Plus T or E for 5 Years | Chemotherapy Plus OFS Plus T or E for 5 Years
Serious Adverse Events (participants affected / at risk) | 0/14 | 6/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OFS Plus T or E for 5 Years (N=14) | Chemotherapy Plus OFS Plus T or E for 5 Years (N=15)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial terminated early due to poor accrual. Adverse event data is available ONLY for selected Grade 3-5 AEs for chemotherapy arm. 25 of 29 patients were co-enrolled in TEXT (IBCSG 25-02), which reports AEs and outcomes of endocrine therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No